CLINICAL TRIAL: NCT05418803
Title: An Open-label, Randomized, 2-sequence, 2-period, Fasted, Single Dose, Oral Administration, Crossover Study to Evaluate the Bioequivalence of YHP1807 Tablets 2.5 mg and YHR1901 Tablets 2.5 mg in Healthy Volunteers
Brief Title: BE Study of Two Formulations of Rivaroxaban 2.5 mg in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHP1807-101
Record Dates: First submitted 2022-06-09; First posted 2022-06-14 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group1 (Experimental): 17 subjects, Cross-over, Single dose of comparator on day1, YHP1807 on day8
  Interventions: Drug: YHP1807 Tab. 2.5mg; Drug: YHR1901 Tab. 2.5mg
- Group2 (Active Comparator): 17 subjects, Cross-over, Single dose of YHP1807 on day1, comparator on day8
  Interventions: Drug: YHP1807 Tab. 2.5mg; Drug: YHR1901 Tab. 2.5mg

INTERVENTIONS:
Drug: YHP1807 Tab. 2.5mg — Rivaroxaban 2.5mg
  Other Names: Experimental
Drug: YHR1901 Tab. 2.5mg — Rivaroxaban 2.5mg
  Other Names: Active comparator

SUMMARY:
The objective of this study was to compare the pharmacokinetic profiles and bioequivalence of rivaroxaban after a single oral dose of rivaroxaban 2.5 mg tablet in healthy Korean subjects.

DETAILED DESCRIPTION:
This study was a randomized, open-label, single-dose, two-period, crossover study which included 34 healthy adult male and female subjects under fasting conditions. A single dose of experimental drug or comparator was administered in each of the two study periods (separated by a washout period of 1 week). Serial blood samples were collected up to 36 hours post-dose. Plasma drug concentrations were measured by liquid chromatography/tandem mass spectrometry (LC-MS/MS). Pharmacokinetic parameters, including maximum plasma concentration (Cmax) and area under the plasma concentration versus time curve from dosing to the last measurable concentration (AUCt), were determined by non-compartmental analysis. The geometric mean ratios and associated 90% confidence intervals (CIs) of log-transformed Cmax and AUCt were calculated to evaluate pharmacokinetic equivalence.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male/female aged 19 to 55 with body mass index(BMI) between 18.5 and 30kg/m2
* Acceptable medical history, physical examination, laboratory tests and EKG, during screening
* Subjects who has signed a written informed consent voluntarily

Exclusion Criteria:

* History of clinically significant medical history or current disease
* Hypotension (SBP ≤ 90 mmHg or DBP ≤ 60 mmHg) or hypertension (SBP

  ≥ 140 mmHg or DBP ≥ 90 mmHg).
* AST(SGOT) or/and ALT(SGPT) > 1.5 times of normal upper limit
* Total bilirubin > 2.0 mg/dl
* Volunteers considered not eligible for the clinical trial by the investigator
* Administration of other investigational products within 6 month prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2020-01-28 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
AUCt | 0-36 hours
  AUCt of Rivaroxaban
Cmax | 0-36 hours
  Cmax of Rivaroxaban

SECONDARY OUTCOMES:
AUCinf | 0-36 hours
  AUCinf of Rivaroxaban
Tmax | 0-36 hours
  Tmax of Rivaroxaban
t1/2 | 0-36 hours
  t1/2 of Rivaroxaban

CONTACTS AND LOCATIONS:
Locations (1):
- Jeonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (including data dictionaries) that underline the results reported in study-related publications will be made available during the period beginning 1 year and ending 5 years after all trial primary and secondary endpoints were assessed. Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to ejsong@yuhan.co.kr.
  A summary of the study results will be posted in the publicly accessible database (i.e. clinicaltrials.gov).
Supporting Information: Study Protocol, CSR
Time Frame: Beginning 1 year and ending 5 years after all trial endpoints were assessed
Access Criteria: Only requests from researchers who provide a methodologically sound proposal will be reviewed and approved by the sponsor. The analysis type should be in accordance with aims in the proposal approved by the sponsor. Proposals should be directed to ejsong@yuhan.co.kr.

REFERENCES:
- [Derived] Moon SJ, Kim Y, Kim SY, Jeon JY, Song E, Lim Y, Kim MG. Comparative pharmacokinetics of two formulations of 2.5-mg rivaroxaban in healthy Korean subjects. Int J Clin Pharmacol Ther. 2023 Mar 5. doi: 10.5414/CP204335. Online ahead of print. PMID 36871246